CLINICAL TRIAL: NCT03938324
Title: Peer i-Coaching for Activated Self-management Optimization in Adolescents and Young Adults With Chronic Conditions
Acronym: PiCASO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00102191; 1R01NR018379-01 (NIH)
Record Dates: First submitted 2019-05-02; First posted 2019-05-06 (Actual); Results first posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Sickle Cell Disease; Chronic Kidney Diseases; Systemic Lupus Erythematosus; Childhood Cancer; Inflammatory Bowel Diseases; Stem Cell Transplant; Organ Transplant; Diabetes Mellitus, Type 1; Cystic Fibrosis
MeSH Terms: conditions — Anemia, Sickle Cell; Renal Insufficiency, Chronic; Lupus Erythematosus, Systemic; Neoplasms; Inflammatory Bowel Diseases; Diabetes Mellitus, Type 1; Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: Five year randomized controlled trial to test efficacy of behavioral intervention versus attention control group on primary and secondary outcomes across 12 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PiCASO Intervention Group (Experimental): Peer coaching intervention delivered by young adults with a childhood onset chronic condition and trained in coaching curriculum that includes motivational interviewing techniques and the benefits of peer relationships over a shared experience such as a chronic condition. The peer coach supports the AYA to identify their goals and feel a sense of success in making change towards goals within a supportive environment. This process involves goal-setting, development of self-discovery and accountability for changes in health behavior. The peer coach elicits the AYA's vision of optimal health and identifies the AYAs values. As the AYAs identify a vision of wellness and develop goals and action steps to progress towards that vision, the peer coach elicits the AYA's intrinsic motivation and activates skill development in self-advocacy and communication and empowers the AYA to take leadership in managing their condition.
  Interventions: Behavioral: PiCASO Intervention Group
- Attention Control Group (Sham Comparator): Over 12 months the attention control group participants will receive a monthly electronic newsletter with educational content about childhood onset chronic condition management and the differences between pediatric and adult health care systems, as well as a monthly phone call from study staff to ensure receipt of the newsletter and to answer questions regarding content, and an opportunity to link them to other resources. If participants report health concerns they will be directed to contact their health care team.
  Interventions: Behavioral: Sham Comparator: Attention Control Group

INTERVENTIONS:
Behavioral: PiCASO Intervention Group — This mobile health intervention utilizes an established telephone/text based secure interface to allow AYAs access knowledge, experience, and instrumental/emotional support from a trained peer coach who has already developed independence an active self-manager. Peers with shared experiences provide instrumental (e.g., health maintenance skills) and emotional support that likely lead to improvements in quality of life. Involving peers in supporting AYAs with chronic conditions to promote self-management and patient activation disrupts the typical over-reliance on the parent and health care provider that often impedes developing independence.
  Arms: PiCASO Intervention Group
Behavioral: Sham Comparator: Attention Control Group — Over 12 months the attention control group participants will receive a monthly electronic newsletter with educational content about childhood onset chronic condition management and the differences between pediatric and adult health care systems, as well as a monthly phone call from study staff to ensure receipt of the newsletter and to answer questions regarding content, and an opportunity to link them to other resources. If participants report health concerns they will be directed to contact their health care team.
  Arms: Attention Control Group

SUMMARY:
The purpose of this study is to test the efficacy of a peer support coaching intervention to improve activated chronic illness self-management versus an attention control group in 225 adolescents and young adults with childhood onset chronic conditions.

DETAILED DESCRIPTION:
Increases in life expectancy in almost all childhood-onset chronic conditions (COCC) has brought unique challenges for adolescents and young adults (AYA) who struggle to deal with the associated disease burden, manage therapies, and thrive as they develop independent self-management skills, and become active and engaged patients. The challenges that influence the lives of AYAs are largely adaptive, such as making lifestyle modifications, adhering to complex medication regimens, and learning to navigate the adult health system. Adding to this complexity is the need for AYAs to progressively take over greater self-management responsibilities from parents. Promoting activated self-management is critically important given that this shift in health care management from parents and health care providers to the AYA is identified as key to successful adult outcomes. Peer support interventions are well-suited to address challenges theorized as critical to AYAs given the importance of peer relationships during this time. The investigators propose a mixed-methods, five-year randomized controlled trial, that will include 225 AYAs (16-22 years) with COCCs, to test the Peer i-Coaching for Activated Self-Management Optimization (PICASO) versus an attention control group. This novel, mobile health intervention utilizes an established telephone/text based secure interface to allow AYAs access knowledge, experience, and instrumental/emotional support from a trained peer coach (18-26 years), who has already developed independence and is an active self-manager. The investigators will determine the efficacy of PICASO on self-management, patient activation, transition readiness, health-related quality, and emotional health of life across 12 months. The investigators will explore whether age, sex, race/ethnicity, chronic condition, and/or disease severity moderate the trajectory of PICASO effects on self-management, patient activation, coping, emotional health and health-related quality of life. Lastly, the investigators will explore mechanisms of the PICASO impact by describing AYA experiences with the intervention.

ELIGIBILITY:
Inclusion Criteria:

* AYA 16 to 22 years
* Childhood onset chronic condition from 1 of 3 condition categories
* Read and speaks English
* Access to internet via computer or Smart Phone
* Access to telephone (Smart Phone not required as text feature can be accessed via internet)

Exclusion Criteria:

* Diagnosed cognitive dysfunction
* Need for English translator

Ages: 16 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Self-representation of gender identity
Enrollment: 222 (Actual)
Dates: Start 2019-10-29 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2024-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angel Barnes, BSN, Study Director — Duke University School of Nursing
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PiCASO Intervention Group | Attention Control Group
Started | 147 | 75
Completed | 99 | 53
Not Completed | 48 | 22
Not completed — Lost to Follow-up | 42 | 21
Not completed — Withdrawal by Subject | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PiCASO Intervention Group | Attention Control Group | Total
Number analyzed (Participants) | 147 | 75 | 222
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.4 (1.9) | 18.3 (1.7) | 18.4 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 45 | 138
  Male | 54 | 30 | 84
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 9 | 22
  Not Hispanic or Latino | 134 | 65 | 199
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 5 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 67 | 20 | 87
  White | 58 | 44 | 102
  More than one race | 4 | 1 | 5
  Unknown or Not Reported | 11 | 7 | 18
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 147 | 75 | 222

OUTCOME MEASURES:

1. Primary Outcome: Change in Self-management as Measured by the Partners in Health Scale
Description: Self-management variable measured using the Partners in Health Scale (PIH): measures chronic illness self-management by assessing chronic condition self-management knowledge, partnership in treatment, recognition and management of symptoms, and coping. This 12 item self-report scale is scored on a 9-point Likert scale. The primary outcome is the overall score, which is the mean of the 12 items (possible range of 0 to 8, higher overall scores indicating better self-management).
Time Frame: baseline, 3, 6, 9, and 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PiCASO Intervention Group | Attention Control Group
Number analyzed (Participants) | 147 | 75
score on a scale
  Baseline | 6.7 (0.7) | 6.5 (0.8)
  3 months | 6.8 (0.7) | 6.6 (0.8)
  6 months | 6.9 (0.8) | 6.6 (0.8)
  9 months | 7.0 (0.8) | 6.6 (0.8)
  12 months | 7.1 (0.8) | 6.6 (0.9)
Statistical Analysis 1: Comparison: PiCASO Intervention Group vs Attention Control Group; Multi-level mixed effects model for longitudinal data to compare treatment group difference in trajectory across 12 months. Group sizes provided at least 80% power to detect a true difference in change trajectories (treatment-by-time interaction effect), assuming a medium effect size, two-tailed tests, and statistical significance set at 0.05. Null hypothesis was no treatment group difference in the trajectory from baseline to 12 months (no significant treatment-by-time effect); Test type: Superiority; p = 0.0034, Multi-level mixed effects — The two-tailed significance set at 0.05 was not adjusted for multiple outcomes or comparisons. No adjustments for pairwise comparisons were required for the model; Fixed effects were treatment, time, treatment-by time; whereas, random effects were participant and participant-by-time

2. Primary Outcome: Patient Activation as Measured by the Patient Activation Measure (PAM-13)
Description: Patient Activation variable measured using the Patient Activation Measure (PAM-13): measures patient activation through self-reports of knowledge, skills, and confidence related to self-management of one's own health care. This 13-item self-report assesses confidence in self-management and understanding of health condition. Each of the 13 items scored on a 5-point Likert scale. The primary outcome is an activation score derived from the 13 items (possible range of 0-100, higher scores indicating higher patient activation in self-management).
Time Frame: baseline, 3, 6, 9, and 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PiCASO Intervention Group | Attention Control Group
Number analyzed (Participants) | 147 | 75
score on a scale
  Baseline | 70.0 (8.4) | 68.8 (8.7)
  3 months | 72.4 (9.2) | 70.8 (9.6)
  6 months | 74.9 (10.0) | 72.8 (10.4)
  9 months | 77.3 (10.9) | 74.8 (11.3)
  12 months | 79.8 (11.7) | 76.8 (12.1)
Statistical Analysis 1: Comparison: PiCASO Intervention Group vs Attention Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.5137, Multi-level mixed effects — [p-value comment as in outcome 1, analysis 1]; Fixed effects were treatment, time, treatment-by time; whereas, random effects were participant and participant-by-time

3. Secondary Outcome: Change in Transition Readiness as Measured by the Transition Readiness Questionnaire (TRAQ 20)
Description: Transition readiness variable measured using Transition Readiness Assessment Questionnaire (TRAQ 20): 20-item self-report assessment of the ability to make appointments, manage medications, track health issues, talk with providers, and manage daily activities. Each item is scored 1-5 on a Likert scale. The primary outcome is the overall score, calculated as the mean of the 20 items (possible range: 1 to 5, higher scores indicating more transition readiness).
Time Frame: baseline, 3, 6, 9, and 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PiCASO Intervention Group | Attention Control Group
Number analyzed (Participants) | 147 | 75
score on a scale
  Baseline | 4.1 (0.5) | 3.9 (0.5)
  3 months | 4.2 (0.4) | 4.0 (0.5)
  6 months | 4.3 (0.4) | 4.1 (0.5)
  9 months | 4.4 (0.4) | 4.1 (0.5)
  12 months | 4.4 (0.4) | 4.2 (0.4)
Statistical Analysis 1: Comparison: PiCASO Intervention Group vs Attention Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.4107, Multi-level mixed effects — [p-value comment as in outcome 1, analysis 1]; Fixed effects were treatment, time, treatment-by time; whereas, random effects were participant and participant-by-time

4. Secondary Outcome: Change in Health-related Quality of Life as Measured by the Short Form Health Survey (SF12) - Mental Component Summary (MCS)
Description: Health-related Quality of Life variable measured using the Short Form Health Survey (SF12): 12-item self-report that assesses health related quality of life. The sum of the MCS items was transformed into T-scores for comparison to the US population (which has a mean of 50 and standard deviation of 10). The MCS T-scores have a range of 0 to 100, with higher scores indicating better mental health status.
Time Frame: baseline, 3, 6, 9, and 12 months
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | PiCASO Intervention Group | Attention Control Group
Number analyzed (Participants) | 147 | 75
T-score
  Baseline | 45.5 (8.1) | 45.1 (8.3)
  3 months | 46.1 (7.8) | 45.1 (8.1)
  6 months | 46.7 (7.5) | 45.1 (7.9)
  9 months | 47.2 (7.3) | 45.1 (7.7)
  12 months | 47.8 (7.2) | 45.1 (7.8)
Statistical Analysis 1: Comparison: PiCASO Intervention Group vs Attention Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.1708, Multi-level mixed effects — [p-value comment as in outcome 1, analysis 1]; Fixed effects were treatment, time, treatment-by time; whereas, random effects were participant and participant-by-time

5. Secondary Outcome: Change in Emotional Health as Measured by the Brief Symptom Inventory (BSI 18)
Description: Emotional health variable measured using the Brief Symptom Inventory: 18-item self-report of emotional symptoms experienced over the previous 7 days. Each item was scored with 0 to 4 Likert scale. The primary outcome was the global severity index score (GSI), an overall score derived by summing the scores of the 18 items (possible range: 0 to 72 with higher scores indicating greater psychological distress).
Time Frame: baseline, 3, 6, 9, and 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PiCASO Intervention Group | Attention Control Group
Number analyzed (Participants) | 147 | 75
score on a scale
  Baseline | 9.7 (8.7) | 10.7 (7.9)
  3 months | 9.5 (9.0) | 10.5 (8.1)
  6 months | 9.3 (9.3) | 10.4 (8.5)
  9 months | 9.0 (9.8) | 10.3 (8.9)
  12 months | 8.8 (10.4) | 10.2 (9.5)
Statistical Analysis 1: Comparison: PiCASO Intervention Group vs Attention Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.7982, Multi-level mixed effects — [p-value comment as in outcome 1, analysis 1]; Fixed effects were treatment, time, treatment-by time; whereas, random effects were participant and participant-by-time

ADVERSE EVENTS:
Time Frame: Up to 12 months
Arm/Group | PiCASO Intervention Group | Attention Control Group
All-Cause Mortality (participants affected / at risk) | 0/147 | 0/75
Serious Adverse Events (participants affected / at risk) | 0/147 | 0/75
Other Adverse Events (participants affected / at risk) | 0/147 | 0/75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-03-11): https://cdn.clinicaltrials.gov/large-docs/24/NCT03938324/Prot_SAP_001.pdf
  • Informed Consent Form (2023-03-24): https://cdn.clinicaltrials.gov/large-docs/24/NCT03938324/ICF_000.pdf